CLINICAL TRIAL: NCT05284643
Title: Pilot Trial of Spectroscopic MRI-guided, Dose-Escalated Proton Radiation Therapy and Bevacizumab for Recurrent Glioblastoma
Brief Title: Spectroscopic MRI, Proton Therapy, and Avastin for Recurrent Glioblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jonathan Bell, Associate Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20210335
Record Dates: First submitted 2022-02-22; First posted 2022-03-17 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Glioblastoma
Keywords: Brain Cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort A: sMRI-Guided RT at 35 Gy in 10 fractions (Experimental): Participants will receive a total dose of 3500 centigrays (cGY) (35Gy) of Spectroscopic Magnetic Resonance Imaging (sMRI)-guided radiation therapy delivered in 10 fractions, 350 cGy (3.5 Gy) to the Clinical Target Volume (CTV) by Intensity Modulated Proton Therapy (IMPT) simultaneous integrated boost technique.
  Participants will also receive Bevacizumab per standard of care, at treating physician's discretion. Initial dose will begin prior to first dose of radiation therapy (RT).
  Interventions: Radiation: Intensity Modulated Proton Therapy (IMPT); Drug: Bevacizumab
- Cohort B: sMRI-Guided RT at 40 Gy in 10 fractions (Experimental): Participants will receive a total dose of 4000 cGY (40Gy) of Spectroscopic Magnetic Resonance Imaging (sMRI)-guided radiation therapy delivered in 10 fractions, 400 cGy (4 Gy) to the Clinical Target Volume (CTV) by Intensity Modulated Proton Therapy (IMPT) simultaneous integrated boost technique.
  Participants will also receive Bevacizumab per standard of care, at treating physician's discretion. Initial dose will begin prior to first dose of radiation therapy (RT).
  Interventions: Radiation: Intensity Modulated Proton Therapy (IMPT); Drug: Bevacizumab

INTERVENTIONS:
Radiation: Intensity Modulated Proton Therapy (IMPT) — Participants will receive radiation therapy delivered via intensity modulated proton therapy (IMPT) simultaneous integrated boost technique over a period of 10 days, 5 days per week for approximately 2 weeks.
Drug: Bevacizumab — Bevacizumab will be administered intravenously (IV), beginning at a dose of 10 mg/kg every 2-3 weeks until disease progression.
  Other Names: Avastin

SUMMARY:
The purpose of this research is to find hidden cancer with an experimental magnetic resonance imaging (MRI) scan called spectroscopic magnetic resonance imaging (sMRI). That spectroscopic MRI scan will be used to increase the area of the brain receiving radiation and then the dose of radiation in attempt to kill more of the cancer. Proton radiotherapy and bevacizumab (Avastin) are used to minimize the possible side effects of this approach.

ELIGIBILITY:
Inclusion Criteria:

A. Recurrent glioblastoma (or variants such as gliosarcoma) based on one of the following criteria:

1. An area of MRI enhancement consistent with glioblastoma outside of the initial high dose radiation field.
2. Biopsy or resection proven recurrent glioblastoma.
3. Progressive glioblastoma based on advanced imaging (brain positron emission tomography (PET), perfusion MRI, or clinical MR Spectroscopy)

B. Pathology diagnosis of glioblastoma, or variants such as gliosarcoma, on initial and/or reresection by 2021 WHO glioblastoma criteria. Prior pathology reports or specimens can be reexamined and reclassified as glioblastoma based on current criteria.

C. Total area of recurrence on T1 post-contrast MRI (including all nodules of likely tumor) have a linear maximum measurement of 6 cm or less.

D. Patients must have received prior brain radiation therapy for glioma in conventional fractionation (1.8 - 2 Gy per fraction, total dose maximum 63 Gy).

E. Patients must have completed prior brain radiation four to six months or more prior to study treatment for recurrent tumors that are at least half based within the high dose (> 46 Gy) radiation field.

1. For "marginal" or "out of field" radiation failures where at least half of the enhancing disease is outside of the prior high dose radiation field but there is field overlap, patients must have completed prior radiation at least four months or more prior to study treatment.
2. For "in field" radiation failures where at least half of the enhancing disease is within the prior high dose radiation field, patients must have completed prior radiation at least six months or more prior to study treatment.

F. A minimum time must be elapsed from the administration of any prior anti-tumor or investigational agents to initiation of study treatments on this protocol as follows:

1. 28 days or 5 half-lives, whichever is shorter, elapsed from the administration of any experimental agent prior to initiation of study treatment.
2. 28 days elapsed from the administration of any prior cytotoxic agents except

i. 14 days from vincristine and ≥ 21 days from procarbazine and Temozolomide (TMZ) prior to initiation of study treatment.

G. Age at least 18.

H. Patients must be able to have MRI scans.

I. Patient must be able to provide written informed consent.

J. ECOG performance status 0-2.

K. Life expectancy greater than 12 weeks at the discretion of the enrolling investigator.qa

L. Female subjects should have a negative serum pregnancy test unless they confirm their menopausal status and/or have undergone previous hysterectomy and/or oophorectomy.

M. Both men and women with childbearing potential should agree to use effective contraception for the duration of the treatment and for at least 6 months after the last treatment since medications that will be used can be harmful for the embryo. See contraception requirements, protocol section 4.16.

N. Complete blood count (CBC)/differential within 21 days prior to registration with absolute neutrophil count at least 1500 cells/mm2, platelets at least 75,000 cells/mm2, and hemoglobin at least 9.0 g/dl (transfusion or other intervention to achieve Hgb of 9.0 or greater is acceptable).

O. Liver function tests must demonstrate total bilirubin 2 mg/dL or less, serum glutamic-oxaloacetic transaminase (SGOT) or aspartate aminotransferase (AST) 2.5 times the upper limit of normal or less within 21 days prior to registration.

P. Kidney function tests must indicate serum creatinine 1.8 mg/dL or less within 21 days prior to registration and the following:

a. Urine protein: creatinine (UPC) ratio < 1.0 within 14 days prior to registration OR urine dipstick for proteinuria ≤ 2+ (patients discovered to have > 2+ proteinuria on dipstick urinalysis at baseline must have a UPC ratio done that is <1.0 to be eligible. If the UPC ratio is ≥ 1.0 then the patients should undergo a 24-hour urine collection and must demonstrate ≤1g of protein in 24 hours to be eligible).

i. Note: UPC ratio of spot urine is an estimation of the 24-hour urine protein excretion; a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm. UPC ratio is calculated using one of the following formulas:

1. [urine protein]/[urine creatinine]: if both protein and creatinine are reported in mg/dL
2. [(urine protein) x0.088]/[urine creatinine]: if urine creatinine is reported in mmol/L

Q. Patients on full-dose anticoagulants must meet both of the following criteria:

1. No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
2. In-range international normalized ratio (INR) (typically 2-3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin, within 21 days prior to registration

Exclusion Criteria:

A. Brain malignancies other than glioblastoma (or variants such as gliosarcoma) by WHO 2021 criteria (benign lesions like meningioma are allowed)

B. Glioma that has not previously undergone standard first line therapies including a first course of radiation therapy.

C. Glioma that has already undergone a second course of radiation therapy.

D. Multi-focal disease (separate enhancing nodules across multiple brain lobes). Note: Multiple nodules in the same region are allowed as long as the total linear diameter is 6 cm or less.

E. Patients who have had treatment with Bevacizumab in the past.

F. Patients who will receive chemotherapy concurrent with study therapy other than bevacizumab.

G. Patients with recurrent Glioblastoma (rGBM) based in the following anatomical regions known to have magnetic susceptibility or poor signal will be excluded: temporal lobe below the level of the floor of the third ventricle, orbitofrontal cortex, prefrontal cortex, medial frontal gyrus, brainstem, and cerebellum (these regions have known sMRI artifact).

H. Pregnant or breastfeeding patients.

I. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1 year. Non-invasive tumors are permissible (e.g., carcinoma in situ).

J. Severe active co-morbidities as follows:

1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration.
2. Transmural myocardial infarction within the last 6 months prior to registration.
3. History of stroke or transient ischemic attack within 6 months prior to registration.
4. Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease.
5. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
6. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
7. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function other than screening panel (Section 3.1) and coagulation parameters are not required for entry into this protocol.
8. Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.

K. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

L. Prior allergic reaction to the study drug (Bevacizumab)

M. Prior history of hypertensive crisis or hypertensive encephalopathy.

N. History of a non-healing wound, ulcer, or bone fracture within 90 days (3 months) prior to registration

O. Gastrointestinal bleeding or any other hemorrhage/bleeding event Common Terminology Criteria for Adverse Events (CTCAE), v. 4 grade 3 or greater within 30 days prior to registration

P. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration (with the exception of craniotomy)

Q. Concurrent receipt of any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients for whom sMRI-guided therapy is technically successful | About 60 days
  The percentage of participants for whom sMRI-guided therapy is successful will be reported as the percentage of participants who show no significant residual tumor after protocol therapy.
Incidence of Grade 3 irreversible or any Grade 4/5 neurologic toxicity. | Up to 6 months
  The incidence of irreversible Grade 3 or any Grade 4/5 neurologic adverse events (AEs) or serious adverse events (SAEs) in study participants will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion. Incidence of these toxicities will be reported for both cohorts, Cohort A (sMRI-Guided RT at 35 Gy in 10 fractions) and Cohort B (sMRI-Guided RT at 40 Gy in 10 fractions).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 2 years
  Progression-free Survival (PFS) is defined as the time from the start of radiation therapy to any documented progression or death from any cause, whichever occurs first. Surviving patients without progression will be censored at the date of last contact.
Overall Survival (OS) | Up to 2 years
  Overall Survival (OS) is defined as the time from the start of radiation therapy to date of death from any cause. Surviving patients will be censored at the date of last contact.
Comparison of Cerebral Blood Volumes (CBV) among MRI techniques | About 3 months
  Comparison of the cerebral blood volumes (CBV) in participants measured by Spectroscopic MRI (sMRI) versus by conventional MRI and multiparametric MRI (mpMRI). CBV is defined as the volume of blood in a given amount of brain tissue, most commonly milliliters of blood per 100 g of brain tissue.
Comparison of Apparent Diffusion Coefficients (ADC) among MRI techniques | About 3 months
  Comparison of the apparent diffusion coefficients (ADC) in participants measured by Spectroscopic MRI (sMRI) versus by conventional MRI and multiparametric MRI (mpMRI). ADC is a measure of the magnitude of diffusion (of water molecules) within tissue, and is commonly clinically calculated using MRI with diffusion-weighted imaging (DWI). ADC of tissue is expressed in units of mm2/s.
Volume of enhancing disease at first progression compared to MRI volumes. | About 3 months
  Assessed by evaluating the patterns of failure after sMRI-guided radiotherapy and correlating with sMRI and other mpMRI markers.
Health-Related Quality of Life (HRQOL) Scores: FACT-Br Questionnaire | Up to 2 years
  Health-Related Quality of Life will be assessed using scores from the Functional Assessment of Cancer Therapy - Brain (FACT-Br) questionnaire version 4. The FACT-Br will be used to evaluate patient function and satisfaction after protocol treatment. The questionnaire has 5 subscales (Physical Well-being, Social/Family Well-being, Emotional Well-being, Function Well-being and Brain Cancer). Response options for each item form a 5-point Likert scale, ranging from 0 ("Not al all") to 4 ("Very Much"). The questionnaire has a total score ranging from 0 - 200, with higher scores representing better HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bell, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No